CLINICAL TRIAL: NCT06093451
Title: An Open-Label, Randomized, Active Controlled Inpatient Trial Evaluating Sublingual Dexmedetomidine For Moderate To Severe Agitation In Inpatients With Schizophrenia Or Bipolar Disorder
Brief Title: Evaluating Sublingual Dexmedetomidine For Moderate To Severe Agitation In Inpatients With Schizophrenia Or Bipolar Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: BioXcel Therapeutics Inc (Industry)
Responsible Party: Principal Investigator, Justin Faden, Associate Professor of Psychiatry, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30561
Record Dates: First submitted 2023-10-05; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia Agitation; Schizo Affective Disorder; Bipolar Disorder; Dexmedetomidine
Keywords: Agitation; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Psychomotor Agitation; Schizophrenia | interventions — Dexmedetomidine; Lorazepam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Participants with moderate agitation will receive sublingual dexmedetomidine 120 mcg as needed. Participants with severe agitation will receive dexmedetomidine 180 mcg as needed.
  Interventions: Drug: Dexmedetomidine
- Lorazapem (Active Comparator): Participants with moderate agitation will receive oral lorazapam 2 mgas needed. Participants with severe agitation will receive oral lorazapam 2 mg as needed.
  Interventions: Drug: Lorazepam 2 MG/ML

INTERVENTIONS:
Drug: Dexmedetomidine — Moderate agitation: 120 mcg Severe agitation: 180 mcg
  Other Names: Igalmi
  Arms: Dexmedetomidine
Drug: Lorazepam 2 MG/ML — 2 mg
  Other Names: Ativan
  Arms: Lorazapem

SUMMARY:
An open-label, randomized, active control inpatient trial to evaluate the efficacy and tolerability of sublingual dexmedetomidine for the treatment of agitation in inpatients with schizophrenia or bipolar disorder as measured by the Positive and Negative Syndrome Scale - Excited Component (PANSS-EC) and Agitation-Calmness Evaluation Scale (ACES). Lorazepam will serve as the active control.

DETAILED DESCRIPTION:
This is an open-label, randomized control trial where patients (N=32) with schizophrenia or bipolar disorder are randomized to receive either sublingual dexmedetomidine or oral lorazepam monotherapy for the treatment of episodic agitation. For moderate agitation (PANSS-EC score ≥14 and <20), patients will receive either sublingual dexmedetomidine 120mcg or oral lorazepam 2mg. For severe agitation (PANSS-EC ≥20), patients will receive either sublingual dexmedetomidine 180mcg or oral lorazepam 2mg. The PANSS-EC and ACES will be evaluated at baseline and after 15, 30, 60, and 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The participant is an adult between the ages of 18-55 at the time of study participation
* Hospitalized on an inpatient unit at Episcopal Hospital
* Meet the DSM-5 criteria for schizophrenia, schizoaffective disorder, or bipolar disorder, as determined by routine clinical assessment conducted upon admission.
* Are able to understand and read English
* Are able to provide informed consent
* Experiencing a moderate (PANSS-EC score ≥14 and <20) or severe (PANSS-EC score ≥20) episode of agitation

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Prisoners
* Participant has an allergy to dexmedetomidine or lorazepam
* Participant has mild, moderate or severe hepatic impairment
* Participant has active pulmonary disease and is receiving treatment (oxygen, inhalers)
* Individual is currently prescribed scheduled benzodiazepines or methadone
* Participant history of QTc ≥ 500 msec or a history of arrythmia
* Participant recent (within the last 2 days) fall, syncope (passing out), feeling lightheaded, or pulse <50.
* Individual has a history of hypokalemia or hypomagnesemia within the past 2 years?
* Participant is receiving high-risk medications, including:

  1. Methadone
  2. Midazolam
  3. Opioids
  4. High risk medications associated with the QT interval prolongation (sertindole, chlorpromazine, ziprasidone), (amiodarone, iboga, quinine, arsenic, ibutilide, selpercatinib, ivosidenib, bedaquiline, lenvatinib, sotalol, levoketoconazole, cisapride, vendetanib, mobocertinib, disopyramide, papaverine)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in PANSS-EC score at 120 minutes after medication administration | Baseline and at 120 minutes
  Severity of agitation will be determined by administering the Positive and Negative Syndrome Scale - Excited Component (PANSS-EC). Moderate to severe agitation will be defined as a PANSS-EC score >=14 and <20; and >= 20 is severe agitation.

SECONDARY OUTCOMES:
Change from baseline in ACES score at 15, 30, 60, 90, and 120 minutes, or prior to receipt of any rescue medication for agitation. | Baseline and 15, 30, 60, 90, and 120 minutes
  Severity of agitation will be measured using the standardized Agitation-Calmness Evaluation Scale. The 9-point scale indicated the degree of agitation as follows: 1=marked agitation, 4=normal behavior, 7 = marked calmness, 9=unarousable.
Change in PANSS-EC score at 15, 30, 60, and 90 minutes, or prior to receipt of any rescue medication for agitation. | Baseline and 15, 30, 60, and 90 minutes
  Severity of agitation will be determined by administering the Positive and Negative Syndrome Scale - Excited Component (PANSS-EC). Moderate to severe agitation will be defined as a PANSS-EC score >=14 and <20; and >= 20 is severe agitation.
Patient tolerability assessed by adverse events of dexmedetomidine | Baseline through 120 minutes after medication administration
  Tolerability and safety of sublingual dexmedetomidine was assessed by evaluating spontaneously-reported adverse events. Treatment tolerability as assessed by adverse events will be tabulated by toxicity grade and organ systems as well as overall.
Patient satisfaction based on Medication Satisfaction Questionnaire (MSQ) | Administered 120 minutes after medication administration
  Medication Satisfaction Questionnaire (MSQ) will be given to the subject to assess their satisfaction of their agitation medication two hours after initial medication administration. The Medication Satisfaction Questionnaire is a 7-point scale, with 1 being "Extremely Dissatisfied", 4 being "Neither Satisfied or Dissatisfied", and 7 being "Extremely Satisfied"
Assess the need for rescue medication for agitation within two hours of medication administration | Baseline and 2 hours after medication administration
  Need for rescue medication of sublingual dexmedetomidine will be assessed by reviewing the Medication Administration Reconciliation (MAR) available on the electronic medical record system for the two hour period of time following medication administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Episcopal Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] San L, Marksteiner J, Zwanzger P, Figuero MA, Romero FT, Kyropoulos G, Peixoto AB, Chirita R, Boldeanu A. State of Acute Agitation at Psychiatric Emergencies in Europe: The STAGE Study. Clin Pract Epidemiol Ment Health. 2016 Oct 27;12:75-86. doi: 10.2174/1745017901612010075. eCollection 2016. PMID 27857778
- [Background] Cots F, Chiarello P, Perez V, Gracia A, Becerra V. Hospital Costs Associated With Agitation in the Acute Care Setting. Psychiatr Serv. 2016 Jan;67(1):124-7. doi: 10.1176/appi.ps.201400508. Epub 2015 Aug 3. PMID 26234333
- [Background] Rubio-Valera M, Luciano JV, Ortiz JM, Salvador-Carulla L, Gracia A, Serrano-Blanco A. Health service use and costs associated with aggressiveness or agitation and containment in adult psychiatric care: a systematic review of the evidence. BMC Psychiatry. 2015 Mar 4;15:35. doi: 10.1186/s12888-015-0417-x. PMID 25881240
- [Background] Richmond JS, Berlin JS, Fishkind AB, Holloman GH Jr, Zeller SL, Wilson MP, Rifai MA, Ng AT. Verbal De-escalation of the Agitated Patient: Consensus Statement of the American Association for Emergency Psychiatry Project BETA De-escalation Workgroup. West J Emerg Med. 2012 Feb;13(1):17-25. doi: 10.5811/westjem.2011.9.6864. PMID 22461917
- [Background] Wilson MP, Pepper D, Currier GW, Holloman GH Jr, Feifel D. The psychopharmacology of agitation: consensus statement of the american association for emergency psychiatry project Beta psychopharmacology workgroup. West J Emerg Med. 2012 Feb;13(1):26-34. doi: 10.5811/westjem.2011.9.6866. PMID 22461918
- [Background] Zeller SL, Citrome L. Managing Agitation Associated with Schizophrenia and Bipolar Disorder in the Emergency Setting. West J Emerg Med. 2016 Mar;17(2):165-72. doi: 10.5811/westjem.2015.12.28763. Epub 2016 Mar 2. PMID 26973742
- [Background] Preskorn SH, Zeller S, Citrome L, Finman J, Goldberg JF, Fava M, Kakar R, De Vivo M, Yocca FD, Risinger R. Effect of Sublingual Dexmedetomidine vs Placebo on Acute Agitation Associated With Bipolar Disorder: A Randomized Clinical Trial. JAMA. 2022 Feb 22;327(8):727-736. doi: 10.1001/jama.2022.0799. PMID 35191924
- [Background] Citrome L, Preskorn SH, Lauriello J, Krystal JH, Kakar R, Finman J, De Vivo M, Yocca FD, Risinger R, Rajachandran L. Sublingual Dexmedetomidine for the Treatment of Acute Agitation in Adults With Schizophrenia or Schizoaffective Disorder: A Randomized Placebo-Controlled Trial. J Clin Psychiatry. 2022 Oct 3;83(6):22m14447. doi: 10.4088/JCP.22m14447. PMID 36198061
- [Background] Igalmi [package insert]. BioXcel Therapeutics, Inc; 2022.